CLINICAL TRIAL: NCT04604470
Title: Trial-specific Patient Decision Aid (tPDA) of the ImmunoSABR Phase 2
Acronym: I-SABR2_PDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: UM2018IMMUNOSABR2RLPL_tPDA
Record Dates: First submitted 2020-10-13; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: NSCLC Stage IV; Lung Cancer; Non Small Cell Lung Cancer; Metastatic Cancer
Keywords: PDA; NSCLC; StageIV; Phase 2 trial; randomized controlled trial; international
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard treatment: Chemotherapy Chemoradiotherapy Radiotherapy Immunotherapy Or a combination of above
  Interventions: Other: Decision tool
- ImmunoSABR treatment: SABR combined immunotherapy
  Radiotherapy combined immunotherapy
  Interventions: Other: Decision tool

INTERVENTIONS:
Other: Decision tool — no intervention.

SUMMARY:
This is a trial-specific (NCT03705403) decision aid (tPDA) for stage IV NSCLC patients that might want to participate.

We want to investigate if a tPDA would be (significantly) helpful for these patients in making a decision.

ImmunoSABR has a complex study design, we expect that the patients get a better overview of the trial via the tPDA because you can bring multiple tools together. (text, video, questions, pictures, timelines, etc.)

DETAILED DESCRIPTION:
A lung cancer patient might want to take part in the ImmunoSABR phase 2 trial (NCT03705403). Before they can decide, it is important that the patients understand why the research is being done and what it would involve for them.

This tPDA will give information about this trial via text, small movies, quiz and preferences. In the end, the patient will receive an overview of their choices.

Detailed Description ImmunoSABR:

IMMUNOSABR will include 126 patients. In this single-stage controlled randomised open-label phase II trial, we aim to demonstrate an absolute increase in progression-free survival (primary endpoint). PFS will be determined as the time between randomisation and disease progression, according to RECIST 1.1, death due to any cause or last patient contact alive and progression-free. Patients will be randomized between control (no immunocytokine) and experimental arms (with immunocytokine L19-IL2) in a 1:1 ratio. The accrual period will be 29 months (or 2.41 years), and the minimum follow-up will be 18 months (or 1.5 years), making the total study duration 47 months. Comparison between control and experimental arms will be made using the Log-Rank statistic. This test for superiority will be one-sided with the desired type I error of 0.10 and power of 0.90.

Patients enrolled in the trial will be randomised into the control arm (C-arm) or experimental arm (E-arm).

C-arm: Standard of Care (SOC) according to the local and national guidelines: (wait and see or surgery and/or chemotherapy and/or standard (symptomatic) radiotherapy and/or SABR, oligometastatic disease.

E-arm: SABR (oligometastatic disease) or radiotherapy (diffuse disease) + L19-IL2 up to 6 cycles (+ aPD(L)1 if SOC) The expected 1.5-year PFS is 15% in the C-arm and 35% in the E-arm. A sample size of 116 patients (58 patients per treatment arm) is needed to show this difference of 20% in PFS, using a logrank test with a two-sided alpha of 0.05 and power of 85%. Patients will be evenly divided over the two arms. Assuming a drop-out rate of 10%, a total of 126 patients (63 per arm) need to be included.

Primary objective The main objective of the trial is to test if the activity of the combination of (SAB)R and L19-IL2 in patients with metastatic NSCLC will result in improved progression-free survival (PFS) compared to the SOC.

Secondary Objectives

Assessment of the PFS of the patient cohort, at 5 years after randomisation. Assessment of the overall survival of the patient cohort, at 5 years after randomisation.

To assess the toxicity of this treatment schedule; To assess Quality of Life (QoL); To assess the occurrence of an Out of Field Radio-Immune (OFRI) response / abscopal effect using imaging; To assess the occurrence of an In Field Radio-Immune (IFRI) response using imaging; To perform correlative biomarker studies related to treatment response.

Exploratory endpoints:

Correlative biomarker studies:

Tumour tissue: e.g EDB expression, non-synonymous mutations, immune monitoring; Blood: e.g. EDB expression, cfDNA, and immune monitoring; Radiomics on CT and if available MRI; Faeces: diversity in microbiota. iRECIST Tumour grow kinetics

ELIGIBILITY:
Inclusion:

Histological confirmed limited metastatic adult NSCLC patients, regardless of the PD-L1 status.

Maximum of 10 metastatic lesions, maximum two brain lesion with a total cumulative diameter of 5cm is allowed.

SOC baseline imaging e.g MRI and/or PET-CT and CT-brain or MRI brain and/or CT-scan with at least covering thorax-upper abdomen-brain, within 6 weeks prior to randomisation.

If a patient has unclear lesions in the liver or brain an MRI would be advised following the ESMO guidelines.

o In patients with 2 lung tumours, it can be unclear if the patient has 2 concurrent primary tumours or a primary lung tumour with 1 metastasis. In this case, the local multidisciplinary tumour board will decide whether the patient has an M1 disease or not.

• Previous treatment: Prior cancer treatments are allowed but must be discontinued for at least 4 weeks before randomisation. In case of maintenance chemotherapy, this therapy will only be started after the end of the L19-IL2 treatment or only in case of Anti-PD(L)1 treatment, during L19-IL2 therapy.

Age of 18 years or older. WHO performance status 0-1; Adequate bone marrow function, evaluated in the local laboratory (Lab): Absolute Neutrophil Count (ANC) of ≥ 1.0 x 109 /L, platelet count ≥ 100 x 109/L, Haemoglobin (Hb) ≥ 6.0 mmol/L (or 9.67 g/dL) (it is allowed to give a blood transfusion if Hb is initially too low); Adequate hepatic function (evaluated in the local lab): total bilirubin ≤ 1.5 x upper limit of normal (ULN) for the institution; ALT, AST, and alkaline phosphatase ≤ 2.5 x ULN for the institution or ≤ 5 in case of liver metastasis); Adequate renal function (evaluated in the local lab): creatinine clearance of at least 40 ml/min; Adequate endocrine (TSH, FT4) function, local guidelines The patient is capable of complying with study procedures; Life expectancy of at least 12 weeks; Negative serum pregnancy test for females of childbearing potential. Signed and dated written informed consent. Ability to comply with contraception requirements

Exclusion criteria

More than 10 metastatic lesions. More than 2 brain metastatic lesions. 2 brain metastases with a cumulative diameter larger than 5 cm. Patients with non-infectious pneumonitis, uncontrolled thyroid disease, pleuritis, pericarditis and peritonitis carcinomatosis.

Patients who received live vaccines 30 days or fewer prior to enrolment. Patients who are already actively participating in another study. Patients who need simultaneous radiation on the primary tumour and metastatic lesion(s). For these patients it might be an option to treat the primary tumour first although this is not mandatory for this study. There must be minimal four weeks between last treatment and randomisation.

Whole brain radiotherapy (WBRT) is not allowed, although it is accepted when given at least 4 weeks prior to randomisation or after the treatment period. Patients with stable brain metastases are not excluded.

Previous radiotherapy to an area that would be re-treated by (SAB)R, resulting in overlap of the high dose areas.

Maintenance therapy with Anti-PD(L)1 treatment combined with chemotherapy is not allowed during treatment ((SAB)R and L19-IL2 cycles).

Other active malignancy or malignancy within the last 2 years (except localised skin basal/squamous cell carcinoma, non-muscle invasive carcinoma of the bladder or in situ carcinoma from any site).

Concomitantly administered glucocorticoids may decrease the activity of IL2 and therefore should be avoided. However, patients who develop life-threatening signs or symptoms may be treated with dexamethasone until toxicity resolves or reduces to an acceptable level (generally grade 1 and 2, however must be based at the research physician's discretion).

History of allergy to intravenously administered proteins/peptides/antibodies/ radiographic contrast media.

HIV positive; active HIV infection, or active hepatitis B or C (assessed in local lab).

Systemic treatment with either corticosteroid (>10 mg daily prednisone equivalents) or Interferon alpha or immunosuppressive medications within 14 days prior to randomisation. Topical or inhalation steroids are allowed. If a patient needs to take unexpectedly immunosuppressive medication during the trial, it will be allowed but decreasing the dose as soon as possible is strongly advised.

Prior history of organ transplant, including autologous stem cell transplant. Acute or sub-acute coronary syndromes within the last year, acute inflammatory heart disease, heart insufficiency NYHA > 2, or irreversible cardiac arrhythmias.

A known impaired cardiac function defined as left ventricular ejection fraction (LVEF) < 50 % (or below the study site's lower limit of normal) as measured by MUGA or ECHO.

Uncontrolled hypertensive disease; (systolic blood pressure (SBP) ≥160 or diastolic blood pressure (DBP) ≥100 mm Hg during two measurements).

History or evidence of active autoimmune disease. Severe diabetic retinopathy (neoangiogenesis targeted by L19 outside the tumour).

Major trauma, including oncologic surgery, but excluding smaller procedures like the placement of porth-à-cath or surgical biopsy, within 4 weeks prior to randomisation (neoangiogenesis targeted by L19 outside a tumour).

Any underlying mental, medical or psychiatric condition which in the opinion of the investigator will make administration of study drug hazardous or hinder the interpretation of study results. Unstable or serious concurrent uncontrolled medical conditions.

Pregnancy or breast feeding; it is well known that ED-B, the target of both L19IL2, is expressed in a variety of fetal tissues. Furthermore, anti-PD(L)1 treatment may increase the risk of immune-mediated disorders. Therefore, it will be contra-indicated for pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Patient's decisional needs to make a decision about participating a clinical trial | 1 year
  Patients' decisional needs (development phase):semi-structured interviews with patients about the decision about their treatment, and what information the patients need to make.
Usability of the decision aid | 1 year
  Quantitative research using a questionnaire based on the International Standard ISO-9242-11. This questionnaire measure to what extent the decision aid is easy to use. Answers will be clear for the patient; agree, neutral, disagree.
Decisional conflict (patients, evaluation phase) | 6months after randomization
  Decisional conflict will be assessed using the DCS (Decisional conflict scale): change in DCS between baseline group (usual care) and ImmunoSABR clinical trial. Answers will be clear for the patient; agree,neutral, disagree. Items are scored and summed. High total score will be in favour of the tPDA
Control Preference Scale (patients; evaluation phase) | 6months after randomization
  Patient's preference to participate in medical decisions will be assessed using the 3-item Control Preference Scale (CPS):change in CPS between baseline group (usual care) and ImmunoSABR clinical trial . Questions and answers will be clear for the patient; agree, neutral, disagree. Items are scored and summed. High total score will be in favour of the tPDA
Perception shared decision-making | 6months after randomization
  Patient's perception of the shared decision-making process will be assessed using the (shared decision making) SDM-Q9 instrument for patients: change in SDM between baseline group (usual care) and ImmunoSABR clinical trial. 9 questions with clear answers; totally disagree, strongly disagree, disagree, agree, strongly agree, totally agree.
Perception shared decision-making | 6months after randomization
  Doctor's perception of the shared decision-making process will be assessed using the SDM-Q9 instrument for professionals: change in SDM between baseline group (usual care) and ImmunoSABR clinical trial. 9 questions with clear answers; totally disagree, strongly disagree, disagree, agree, strongly agree, totally agree.

SECONDARY OUTCOMES:
Patients' satisfaction with decision aid | 6months after randomization
  Patients satisfaction with the tPDA will be tested via questions with predefined answers; agree,neutral, disagree. Items are scored and summed. High total score will be in favour of the tPDA
Patients' intention to use and recommend tPDA to others | 6months after randomization
  Patients recommendation regarding the tPDA will be tested via questions with predefined answers; agree, neutral, disagree. Items are scored and summed. High total score will be in favour of the tPDA

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, Prof. MD, Study Director — MUMC/UM

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of ImmunoSABR trial — https://www.immunosabr.info/
- See also: Page of ImmunoSABR phase 2 trial on Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT03705403